CLINICAL TRIAL: NCT05914480
Title: Sepsis in ICU: Causes and Outcomes in Diabetics and Non Diabetics in Assiut University Hospital
Brief Title: Sepsis in ICU:Causes and Outcomes in Diabetics and Non Diabetics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Ahmed fathi mansour, Specialist, Assiut University
Other Study IDs: Sepsis pts investigate causes
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PCR for legionella ,blood ,urine cultures and from catheters or source of infection — Investigations to detect cause of sepsis as blood cultures ,urine cultures and from catheters .also PCR for legionella will be done

SUMMARY:
Identify prevalence of sepsis in ICU of Assiut university hospital 2.Clarify different causes of sepsis in patients admitted to ICU . 3.Compare causes and outcomes of sepsis between diabetics versus non diabetics .

4.Screening for the co1.mmonest organism causing sepsis in critically ill patients .

DETAILED DESCRIPTION:
Sepsis, is defined as an infection with organ dysfunction, There is wide variation in sepsis rates, causative microorganisms, and outcome in ICU patients around the world.

Many conservative estimates considered sepsis as a leading cause of mortality and critical illness worldwide .

sepsis epidemiology studies worldwide revealed a highly variable incidence of 13-300 per 100,000 inhabitants per year for severe sepsis and 11 per 100,000 inhabitants per year for septic shock .

Factors such as advancing age, immunosuppression and multidrug-resistant infection play a role in increasing incidence of sepsis during recent decades .

Patients who survive sepsis often have long-term physical, psychological, and cognitive disabilities with significant health and social implications.

Patients with diabetes mellitus have an increased risk of developing infections and sepsis and they constitute 20.1-22.7% of all sepsis patients.

The prevalence of diabetes mellitus in ICU patients is as high as 30%, And such patients are at increased risk of experiencing in-hospital Complications, compared to patients without diabetes.

Infective complications may be reduced with lower blood glucose concentrations Moreover, in critically ill patients without diabetes, Hyperglycemia is associated with increased mortality, risk of infection, Kidney injury and cardiovascular complications.

Moreover, diabetes is a major risk factor for both Acute Kidney Injury and sepsis.

Sepsis also is a major cause of Acute Kidney Injury, which develops in one-fourth of all patients with sepsis and half of patients with bacteraemia or shock .

Sepsis-related AKI is associated with high mortality rates of up to 70%.

ELIGIBILITY:
Inclusion Criteria:

* according to sofa criteria Suspected /documented infection+sofa score >_2 or +ve Q sofa defined as 2or more 1_ hypotesion SBP<90.2_altered mental status GCS<13 3_ Exclusion Criteria:tachypnea>22 or septic shock criteria
* previous history of pulmonary problem Previous history of cardiac disease Previous history of autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ICU diagnosed as sepsis or septic shock even on admission or later on then subdivided into 2 groups 1_Hyperglycemic (diabetic and non diabetic) .2_Normoglycemic(diabetic and non diabetic)
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Detect the most common organism causing sepsis in ICU | 20 days
  Applying culture and sensitivity test for patients developed sepsis on admission and follow up will direct us for appropriate treatment for all patients

SECONDARY OUTCOMES:
Incidence of sepsis in diabetics versus non diabetics in ICU. | 15 days
  Assess the effect of hyperglycemia on spsis outcomes.